CLINICAL TRIAL: NCT07365644
Title: Prophylactic ANTicoagulation With HEparine in Critically Ill Patients With Renal Impairment
Acronym: PANTHER
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2025/S03/14
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Prophylactic Anticoagulation
Keywords: intensive care unit; Prophylactic ANTicoagulation; Renal impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with impaired renal function in intensive care

SUMMARY:
Intensive care patients have an increased risk of venous thromboembolic events (deep vein thrombosis (DVT) and pulmonary embolism (PE)) due to the presence of general risk factors for thrombosis (age, immobilization, obesity, prothrombotic history, etc.), but also risk factors specifically related to their stay in intensive care (sepsis, vasopressors, organ failure, mechanical ventilation, sedation, renal failure, central venous catheters). In addition, these same patients also have an increased risk of hemorrhagic events, mainly associated with coagulation disorders and thrombocytopenia.

Given this increased risk of thrombosis, it is recommended that heparin thromboprophylaxis be used in intensive care patients in the absence of contraindications.

In current practice, when faced with a patient with impaired renal function, there is significant heterogeneity in the prescription of thromboprophylaxis between centers and intensive care physicians: some will use enoxaparin, dalteparin, or tinzaparin regardless of renal function, while others will use subcutaneous calciparin or IVSE UFH.

The PANTHER study is a prospective, multicenter, observational study that aims to evaluate the safety and efficacy of heparin thromboprophylaxis in critically ill patients with renal failure. The goal is to assess whether there is a difference in bleeding risk and thromboprophylaxis efficacy depending on the molecule used.

ELIGIBILITY:
Inclusion Criteria:

* Presence of impaired renal function (one of the two criteria must be met, both criteria may be met):

Glomerular filtration rate (GFR) <30ml/min/1.7m² according to the MDRD or CKD-EPI formula.

Acute renal failure (observed or presumed increase in creatinine in the last 7 days) KDIGO stage 3 (creatinine ≥3 times baseline creatinine or ≥354 µmol/L (4 mg/dL) or urine output <0.3 mL/kg/h for ≥24 hours or initiation of extrarenal clearance or anuria for ≥12 hours)

- Expected length of stay in intensive care ≥48 hours

Exclusion Criteria:

* Age ≤ 18 years
* Long-term dialysis patient
* Current or recent hemorrhage during this hospitalization
* Patient receiving curative anticoagulation or treated long-term prior to admission with curative anticoagulation.
* Thrombosis present on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with impaired renal function in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 1111 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of hemorrhagic and thrombotic events in patients with renal failure in intensive care receiving heparin thromboprophylaxis | Day 1 to Day 28
  Incidence of hemorrhagic and thrombotic events was evaluated by occurrence of major bleeding and occurrence of a venous thromboembolic event

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU Angers, Angers
  - CHU bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Caen, Caen
  - Centre Hospitalier Le Mans, Le Mans
  - Groupe Hospitalier Bretagne Sud, Lorient
  - CHR Metz-Thionville site Mercy, Metz
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Orléans, Orléans
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - Centre Hospitalier de Saint-Nazaire, Saint-Nazaire
  - CHR Metz-Thionville Hôpital Bel-Air, Thionville
  - CHU Tours, Tours